CLINICAL TRIAL: NCT04208555
Title: A Randomized Comparison of Boric Acid Versus Terconazole in Treatment of Recurrent Vulvovaginal Candidiasis
Brief Title: Comparison of Boric Acid vs. Terconazole in Treatment of RVVC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hatem AbuHashim (Other)
Responsible Party: Sponsor-Investigator, Hatem AbuHashim, Professor, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS.19.09.825
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Vulvovaginal Candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Boric acid vaginal suppository (Experimental)
  Interventions: Drug: Boric Acid Vaginal Suppository
- Terconazole vaginal suppository (Active Comparator)
  Interventions: Drug: Terconazole Vaginal Suppository

INTERVENTIONS:
Drug: Boric Acid Vaginal Suppository — Boric acid vaginal suppository (600 mg/day) for 14 days
  Arms: Boric acid vaginal suppository
Drug: Terconazole Vaginal Suppository — Terconazole 80 mg vaginal suppository daily for 6 days
  Arms: Terconazole vaginal suppository

SUMMARY:
Vulvovaginal candidiasis (VVC) caused by Candida species, predominantly C. Albicans is considered one of the most common infections of the lower female genital tract affecting 75% of women at least once in their lifetime. Recurrent VVC (RVVC) is arbitrarily defined as four or more episodes every year. RVVC is a debilitating, long-term condition that can severely affect the quality of life of women. Several factors have been associated with RVVC such as prolonged use of antibiotics, inadequately treated infection, uncontrolled diabetes, immune mechanisms (e.g. HIV), oral contraceptive use as well as the resistance of non-albicans Candida species (e.g. C glabrata, C krusei) to conventional antifungal agents as azoles.

Fluconazole administered orally is the most commonly used antifungal drug in the case of RVVC. However, in the last decade, fluconazole-resistant C Albicans has been reported in women with RVVC. Terconazole is a broad-spectrum, triazole antifungal treatment agent for both C Albicans and non-albicans. Its use (80 mg vaginal suppository daily for 6 days) was as effective as two doses of oral fluconazole (150 mg) in the treatment of patients with severe VVC and RVVC.

Boric acid or boracic [B(OH)3] is a weak acid with proven antifungal action. In RVVC especially in azole-resistant strains and in non-Candida Albicans, 600 mg of the boric acid vaginal suppository is recommended once daily for 2 weeks. This regimen has a mycologic cure rate varied from 40% to 100%. However, there are no published studies comparing the intravaginal use of boric acid with terconazole for RVVC. Accordingly, a prospective randomized study in patients with RVVC will be conducted to address this important issue.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RVVC will be defined as four or more episodes of VVC that occurred during the previous 12-month period.
* Has symptoms and signs of VVC e.g. itching, burning, discharge, and erythema.
* Documented VVC on high vaginal swabs (HVSs) by the demonstration of blastospores and pseudohyphae in a wet vaginal smear treated with 10% potassium hydroxide, and a positive fungal culture.
* Age: 18-50 years old and premenopausal.
* Agree to abstain from sexual intercourse during the treatment period.
* Agree to abstain from using any other vaginal product during the study period.

Exclusion Criteria:

* Postmenopausal.
* Pregnancy.
* Sexually transmitted infection (Chlamydia, gonorrhea, trichomonas).
* Any antifungal or antibiotic use 14 days prior to treatment.
* Gynecological conditions requiring treatment e.g. Bartholin's cyst, abscess, PID.
* Patients receiving corticosteroids or immunosuppressive therapy.
* Patients expected to menstruate within seven days of the start of treatment.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2020-01-15 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Mycological cure rate | At day 15 of treatment
  Negative Candida by cultures of high vaginal swabs

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Abu Hashim, MD. FRCOG. PhD, Study Chair — Faculty of Medicine, Mansoura University; Asmaa Swidan, MBBCh, Principal Investigator — New Mansoura General Hospital

REFERENCES:
- [Background] Iavazzo C, Gkegkes ID, Zarkada IM, Falagas ME. Boric acid for recurrent vulvovaginal candidiasis: the clinical evidence. J Womens Health (Larchmt). 2011 Aug;20(8):1245-55. doi: 10.1089/jwh.2010.2708. Epub 2011 Jul 20. PMID 21774671